CLINICAL TRIAL: NCT06185556
Title: COLDFIRE-III Trial: Perivascular and Peribiliary Colorectal Liver Metastases (0-5cm): Irreversible Electroporation Versus Stereotactic Body Radiotherapy
Brief Title: COLDFIRE-III Trial: Efficacy of Irreversible Electroporation and Stereotactic Body Radiotherapy for Perivascular and Peribiliary Colorectal Liver Metastases
Acronym: COLDFIRE-III
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Angiodynamics, Inc. (Industry)
Responsible Party: Principal Investigator, M.R. Meijerink, Prof. dr., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL83557.018.23
Record Dates: First submitted 2023-11-17; First posted 2023-12-29 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer; Liver Metastases; Liver Metastasis Colon Cancer; Unresectable Solid Tumor
Keywords: Colorectal liver metastases; colorectal hepatic metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Electroporation; Radiosurgery

STUDY DESIGN:
Intervention Model Description: A prospective, randomized clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: Irreversible electroporation (Active Comparator): Irreversible electroporation (IRE) is a primarily non-thermal, local ablative technique that utilizes electrical pulses to destroy tumor tissue. Theoretically, IRE only affects viable tumor tissue, leaving surrounding vital structures relatively intact. It is therefore considered to cause less morbidity than thermal ablative strategies.
  Interventions: Procedure: Irreversible electroporation
- B: Stereotactic body radiotherapy (Active Comparator): Stereotactic body radiotherapy (SBRT) is a form of external beam radiation that has important advantages over conventional radiotherapy such as a more precise and greater biological dose delivery and hence less toxicity and presumably better outcome.
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Procedure: Irreversible electroporation — Percutaneous (CT-guided) irreversible electroporation of 1-3 perivascular and peribiliary colorectal liver metastasis.
  Arms: A: Irreversible electroporation
Radiation: Stereotactic body radiotherapy — Stereotactic body radiotherapy (CT- or MRI-guided) of 1-3 perivascular and peribiliary colorectal liver metastases.
  Arms: B: Stereotactic body radiotherapy

SUMMARY:
The primary objective of this phase IIb/III, prospective, randomized clinical trial is to compare the efficacy of irreversible electroporation (IRE) with stereotactic body radiotherapy (SBRT) in patients with perivascular or peribiliary colorectal liver metastases (CRLM), that are not amenable for surgical resection or thermal ablation. Efficacy is assessed in terms of local control at 2 years.

DETAILED DESCRIPTION:
Rationale: Currently, the gold standard for perivascular and peribiliary colorectal liver metastases (CRLM), that are not amenable for surgical resection or thermal ablation, is undetermined. Two non-thermal treatment modalities could provide a solution for these anatomically challenging CRLM: irreversible electroporation (IRE) and stereotactic body radiotherapy (SBRT).

IRE is a new, minimal-invasive image-guided treatment method for tumors not amenable for surgical resection or thermal ablation, due to vicinity near vital structures such as vessels and bile ducts. With IRE, multiple electrical pulses are applied to tumorous tissue. These pulses alter the existing transmembrane potential of the cell membranes, and create 'nanopores', after which the cell dies through loss of homeastasis. SBRT is another non-thermal ablation modality and has important advantages over conventional radiotherapy such as a more precise and greater biological dose delivery and hence less toxicity and presumably better outcome.

Study design: The COLDFIRE-III trial is a phase IIB/III, prospective randomized clinical trial. The primary conducting center will be the Amsterdam UMC (Amsterdam, the Netherlands). The purpose of this study is to assess and compare the efficacy of IRE and SBRT for perivascular or peribiliary CRLM in terms of local control at 2 years. Other objectives are overall survival, additional efficacy endpoints, safety, pain assessments and costs. For the sample size calculations, the log-rank test is used. The (2-year survival) proportion in group 1 (a treatment group) is 0.80. The proportion in group 2 (the alternative treatment group) is 0.55. The significance level of the test is 0.10. A total number of 78 patients will be randomized into one of two arms: arm A (IRE, n = 39) and arm B (SBRT, n = 39).

Study population: 78 patients with 1-3 perivascular and peribiliary lesions of 0-5 cm, ineligible for surgical resection and thermal ablation, suitable for both IRE and SBRT and no or limited extrahepatic disease (1 extrahepatic lesion is allowed, not including positive para-aortic lymph nodes, celiac lymph nodes, adrenal metastases, pleural carcinomatosis or peritoneal carcinomatosis) can be included. Supplementary resections for resectable lesions and thermal ablations for unresectable CRLM are allowed. A maximum number of 10 CRLM are allowed for patients with no extrahepatic disease and a maximum number of 5 lesions are allowed for patients with limited extrahepatic disease. Eligible patients will be stratified according to tumor size (≤3cm vs. 3-5 cm) and (induction) chemotherapy prior to local treatment.

Intervention: Patients will be randomized into one of two arms, arm A (IRE) and arm B (SBRT). The expert panel, consisting of at least two interventional radiologists, two radiation oncologists and two hepatobiliary surgeons, will appoint lesions that are ineligible for surgery of thermal ablation, and suitable for both IRE and SBRT, as target lesions.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of primary colorectal tumor is available;
* 1-3 CRLM visible on ceCT and/or MRI, size 0-5 cm and not eligible for resection or thermal ablation due to location close to a vessel or bile duct;
* Additional CRLM are allowed if considered either resectable or ablatable with a maximum of 10 CRLM. In patients with extrahepatic disease, a maximum of 5 additional CRLM is allowed;
* No or limited extrahepatic disease (1 extrahepatic lesion is allowed, with some exclusions mentioned in the exclusion criteria);
* Prior focal liver treatment is allowed;
* Subjects should preferably be treated with neo-adjuvant systemic therapy;
* Subjects with recurrent (either local or distant-hepatic) CRLM after previous focal treatment who are unsuitable for (further) systemic therapy (further downsizing or conversion to resectable disease improbable);
* Adequate bone marrow, liver and renal function as assessed by laboratory requirements to be conducted within 7 days prior to definite inclusion;
* ASA classification 0 - 3;
* Age >18 years;
* Written informed consent;

Exclusion Criteria:

* Radical treatment unfeasible or unsafe (e.g. insufficient FLR);
* >10 CRLM; >5 CRLM when extra-hepatic disease is present;
* Positive para-aortal lymph nodes, celiac lymph nodes, adrenal metastases, pleural carcinomatosis or peritoneal carcinomatosis;
* Subjects who have progressive disease after neo-adjuvant systemic therapy;
* History of epilepsy;
* History of cardiac disease:
* Uncontrolled hypertension. Blood pressure must be ≤160/95 mmHg at the time of screening on a stable antihypertensive regimen;
* Compromised liver function (e.g. signs of portal hypertension, INR > 1,5 without use of anticoagulants, ascites);
* Pregnant or breast-feeding subjects;
* Immunotherapy ≤ 2 weeks prior to the procedure;
* Chemotherapy and/or targeted therapy ≤ 2 weeks prior to the procedure;
* Severe allergy to contrast media not controlled with premedication;
* Any condition that is unstable or that could jeopardize the safety of the subject and their compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Local control | 2 years
  Local control is defined as no objectified signs for local tumor progression on imaging acquired 23-24 months following start of the initial study procedure, according to the RECIST criteria. Site recurrences within the first 12 months that are successfully retreated once using the same technique (re-IRE or re-SBRT), thermal ablation or surgical resection will not be regarded as an event for local control. Per patient analysis.

SECONDARY OUTCOMES:
Overall survival (OS) per patient | Assessed up to 5 years
  Overall survival is defined as the time from randomization to the time of death due to any cause or to the last day of follow up (censored).
Local tumor progression-free survival (LTPFS) per patient and per tumor. | Assessed up to 5 years
  Local tumor progression-free survival is defined as the time from randomization to the time of unequivocal local tumor progression.
Distant tumor progression-free survival (DPFS) per patient | Assessed up to 5 years
  Distant tumor progression-free survival is defined as the time from randomization to the time of unequivocal distant tumor progression.
Time to progression (TTP) per patient | Assessed up to 5 years
  Time to progression is defined as the time from randomization to the time of local disease progression, new metastases (events). The date of death from any cause is considered to be a competing risk
Safety per procedure and per patient | Assessed up to 5 years
  Rate of adverse events and serious adverse event, graded from I to V according to the standard classification of surgical complications.
Assessment of pain per patient | Assessed up to 1 year
  Pain assessment using visual analogue scale questionnaires (VAS; per procedure analysis: Assessed prior to, directly after and every three months after local treatment.
Quality of life (QoL) per patient as assessed by EORCT QLQ-C30 questionnaires | Assessed up to 1 year
  The quality of life is assessed in both treatments using EORCT QLQ-C30 questionnaire (per procedure analysis), prior to, and every three months after treatment during a total follow-up time of 1 year.questionnaires: Assessed prior to, and every three months after local treatment.
Quality of life (QoL) per patient as assessed by EQ-5D questionnaires | Assessed up to 1 year
  The quality of life is assessed in both treatments using EQ-5D questionnaire (per procedure analysis), prior to, and every three months after treatment during a total follow-up time of 1 year.questionnaires: Assessed prior to, and every three months after local treatment.
Quality of life (QoL) per patient as assessed by PRODISQ questionnaires | Assessed up to 1 year
  The quality of life is assessed in both treatments using PRODISQ questionnaire (per procedure analysis), prior to, and every three months after treatment during a total follow-up time of 1 year.questionnaires: Assessed prior to, and every three months after local treatment.
Cost-effectiveness ratio (ICER) per patient | Assessed up to 5 years
  Direct and indirect total costs of care, and incremental cost-effectiveness ratio (ICER).

CONTACTS AND LOCATIONS:
Overall Officials: Martijn R. Meijerink, Prof., Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC - location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No